CLINICAL TRIAL: NCT05312320
Title: Improving Sexual Function After Myocardial Infarction - a Randomized Controlled Trial.
Brief Title: Improving Sexual Function After Myocardial Infarction
Acronym: Sex/MI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20/09003-10-521
Record Dates: First submitted 2022-03-11; First posted 2022-04-05 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-03

CONDITIONS: Sexual Function Disturbances; Myocardial Infarction
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Information film (Active Comparator): Randomized to receive a short information film online.
  Interventions: Other: Information film
- Standard care (No Intervention): No film, only questionnaire.

INTERVENTIONS:
Other: Information film — * Sexual activity after MI does not increase risk of recurrence or death
  * Sexual activity is associated with improved outcome after MI
  * Resuming sexual activity as normal is recommended and completely safe
  Arms: Information film

SUMMARY:
The study is completely digital. Men and women who recently had an MI will be invited through a written brochure that will be present in all Norwegian departments of cardiology. Post-MI patients can check the investigators web site (www.sefh.no) to determine whether they are eligible for the study. After consent and answering the baseline questionnaire, each participant will be randomized to either the intervention or control group.

Control group: Standard surveillance after MI (no specific focus on sexual activity and functioning) Intervention group: Online sexual counselling including a short information film.

In order to assess the generalizability of the results, we will compare the age, sex and MI treatment of the respondents with data on Norwegian MI-patients in general.

DETAILED DESCRIPTION:
The investigators will include 600 women and 600 men within 4 weeks after an acute MI. The investigators will invite the same number of women and men from the general population, invited through mass and social media.

All participants will be provided the same questionnaire at 4 weeks. Then outcome data will be obtained by a follow-up quest after 6 and 12 months.

The intervention is a film with the following main message:

* Sexual activity after MI does not increase risk of recurrence or death
* Sexual activity is associated with improved outcome after MI
* Resuming sexual activity as normal is recommended and completely safe

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years old
* Acute MI during the last 6 weeks
* Informed consent for participation

Exclusion Criteria:

* Lack of ability to cooperate
* Known alcohol- or drug-abuse, or use of narcotics
* Pregnancy or breast-feeding
* Serious comorbidity with a life expectancy <12 months
* Unstable or refractory angina
* Uncontrolled hypertension
* Congestive heart failure (NYHA class III/IV)
* High-risk arrhythmias
* Hypertrophic obstructive and other cardiomyopathies
* Severe valvular disease

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Does specific sexual counselling improve sexual functioning in post-MI? | 12 months
  The investigators will measure sexual function by Brief Sexual Function Inventory (BSFI) for male participants and Female Sexual Function Index (FSFI) for female participants at 6 and 12 months after their MI.
Changes in sexual activity and functioning after MI | 12 months
  The investigators will measure sexual activity and function at baseline, and 6 and 12 months after MI.
  The investigators will measure sexual function by Brief Sexual Function Inventory (BSFI) for male participants and Female Sexual Function Index (FSFI) for female participants.
Establish predictors of improved sexual functioning in post-MI patients | 12 months
  In order to identify MI patients at risk of sexual dysfunction, the participants will answer questionnaires on quality of life (RAND-12), depression and anxiety (HADS), demographic data, comorbidity, medications and other factors that may have impact on sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Frode Gallefoss, Study Director — Sorlandets hospital HF
Locations (1):
- Www.Sefh.No, Arendal, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: control group — http://betami.org